CLINICAL TRIAL: NCT03052543
Title: A Pilot Study to Determine the Outcomes of an Intraoperative Bispectral Index Monitor
Brief Title: Outcomes of an Intraoperative Bispectral Index Monitor
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Keira Mason, principal investigator, Boston Children's Hospital
Other Study IDs: IRB-P00024412
Record Dates: First submitted 2017-01-03; First posted 2017-02-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- BISblind: The BISblind group will have the BIS monitor and data physically hidden from the anesthesiologist. The patient will receive an anesthetic as per the anesthesiologist's particular care plan, unaltered by the study.
  Interventions: Device: BIS™ Complete 2--Channel Monitor
- BISvisible: BISvisible group will have the BIS monitor and data available for the anesthesiologist to view. The patient will receive an anesthetic as per the anesthesiologist's particular care plan, unaltered by the study.
  Interventions: Device: BIS™ Complete 2--Channel Monitor

INTERVENTIONS:
Device: BIS™ Complete 2--Channel Monitor — monitor depth of anesthesia

SUMMARY:
This pilot study is being conducted to determine whether the intraoperative presence of a Bispectral Index Monitor (BIS), a non-invasive monitor, affects the perioperative and postoperative indices and outcomes. The BIS monitor is an adhesive sensor that is applied to the forehead to monitor EEG waves. This monitor is not a Standard of Care Monitor, yet in adult and pediatric studies it has been shown to decrease time to emergence, decrease volatile anesthesia requirement, decrease recovery time and in some cases, decrease post-operative morbidity (REFS). The effect on intra-operative and post-operative parameters, when BIS is present but not specifically designated to be used as a monitor to guide anesthesia delivery, has not been specifically examined. This will be the first pediatric study which applies BIS on all patients and randomizes the anesthesiologists to either be or not be privy to seeing the BIS values during intra-operative period.

DETAILED DESCRIPTION:
The BIS monitor is an adhesive sensor that is applied to the forehead to monitor EEG waves. In adult and pediatric studies, the BIS monitor has been shown to decrease time to emergence, decrease volatile anesthesia requirement, decrease recovery time and in some cases, decrease post-operative morbidity (REFS). The effect on intra-operative and post-operative parameters, when BIS is present but not specifically designated to be used as a monitor to guide anesthesia delivery, has not been specifically examined. This will be the first pediatric study which applies BIS on all patients and randomizes the anesthesiologists to either be or not be privy to seeing the BIS values during intra-operative period.

ELIGIBILITY:
Inclusion Criteria:

* orthopedic or urologic day surgery
* 2 to 12 years old

Exclusion Criteria:

* anesthesiologist refusal
* patient/parent refusal
* allergy to the BIS adhesive
* history of seizures

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 60 patients ages 2-12 scheduled for day surgery at Boston Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
BIS values | intraoperative period
  Compare the BIS values in the BISblind and BISvisible groups

SECONDARY OUTCOMES:
Amount of intravenous anesthetic medications administered | intraoperative period
  Compare the amount of intravenous anesthetic medications administered between the BISblind and BISvisible groups
End tidal sevoflurane values | intraoperative period
  Compare the end tidal sevoflurane values between the BISblind and BISvisible groups
Agitation/delirium | post operative period, until discharge from recovery room, assessed up to 10 hours
  Determine the incidence of agitation and delirium using the post-anesthesia emergence delirium scale in the post anesthesia care unit
Pain scores | post operative period, until discharge from recovery room, assessed up to 10 hours
  Compare the pain scores between the BISblind and BISvisible groups
Time to meet discharge criteria | post operative period, until discharge from recovery room, assessed up to 10 hours
  Compare the time needed to meet discharge criteria between the BISblind and BISvisible groups

CONTACTS AND LOCATIONS:
Overall Officials: Keira Mason, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No